CLINICAL TRIAL: NCT07350148
Title: Integrating Mindfulness and mHealth Approaches for Treating Opioid Use Disorder
Brief Title: Opioid Adherence and Support Through Innovative Texting Strategies
Acronym: OASIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2507214546; K23DA058015 (NIH)
Record Dates: First submitted 2026-01-14; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder (OUD); Chronic Pain
Keywords: text message; medications for opioid use disorder; mHealth; mindfulness; medication adherence
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain; Medication Adherence

STUDY DESIGN:
Intervention Model Description: The study uses a micro-randomized trial design which randomizes the number of mindfulness text messages sent to each participant each day.
Masking Description: All data are collected online, without the research team's involvement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness text messages (Experimental)
  Interventions: Behavioral: Mindfulness text messages

INTERVENTIONS:
Behavioral: Mindfulness text messages — Over 250 text messages based on concepts from Mindfulness-Based Relapse Prevention (MBRP) were developed and are sent to participants each day for 4 weeks. The messages are intended to increase awareness of triggers and "automatic" reactions to triggering experiences, and to consider alternative responses to these experiences.

SUMMARY:
The goal of this clinical trial is to examine the effects of reminder and mindfulness text messages on medication adherence and managing craving, pain, and withdrawal symptoms in people taking medications for opioid use disorder through assessment questions collected twice daily during the course of treatment. The main questions it aims to answer are:

1. Do daily medication reminder text messages increase medication adherence for people taking medications for opioid use disorder?
2. To what extent do people engage with the daily mindfulness messages?
3. What impact does daily mindfulness text message quantity have on craving, pain, forgetfulness, and withdrawal symptoms?

Participants will:

1. Receive daily medication reminder text messages for at least 24 weeks (i.e., 6 months)
2. Receive up to 6 mindfulness messages per day for 4 weeks (i.e., 1 month)
3. Answer daily questions twice a day during the 4 weeks of mindfulness messages
4. Answer questions about the study when enrolling, at the end of the 4 weeks of mindfulness messages, and at 4 and 16 weeks after the end of the mindfulness messages

DETAILED DESCRIPTION:
This study will examine the acceptability, feasibility, and effectiveness of mindfulness text messages in increasing adherence to medications for opioid use disorder and in helping people manage pain, craving, and withdrawal symptoms. The study sends up to six daily mindfulness text messages for 4 weeks as well as daily medication reminder text messages for at least 24 weeks. The study uses a micro-randomized trial design and participants are randomized each day to receive a random number of mindfulness messages (range: 0 to 6). The investigators will compare self-reported daily medication adherence to typical rates reported in the literature. Additionally, the study will examine the impact of text message quantity on primary constructs of interest (craving, pain/pain interference, withdrawal symptoms). Secondary constructs of interest collected during the mindfulness texting period include message engagement, state mindfulness, state values-based living, substance misuse, and self-efficacy. People (n=60) who report initiating or restarting taking daily medication for opioid use disorder (e.g., methadone, buprenorphine/suboxone/subutex) will be enrolled in the study. Participants will answer questions about their functioning, mood, quality of life, sleep, substance use, pain, and more at baseline, and at follow-up months 1, 2, and 6 (4, 8, and 24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have a cellphone that can receive text messages
* Have internet access to complete study surveys
* Willing to comply with all study procedures and be available for the duration of the study
* Within 6 months of starting or resuming to take daily methadone or buprenorphine (or suboxone/subutex)
* Able to understand study requirements and provide informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Mindfulness text intervention engagement | Measured daily for four weeks
  Participants reply to a binary ("Today, did you think about or use any suggestion from the OASIS Study text messages?") and continuous ("How much did you think about or use any suggestion from the OASIS text messages?; response range: 0=not at all, 10=very much) question about intervention engagement. They also indicate how much they believe the texting helped them manage their pain, urge to use opioids, remember to take their medication, and manage their withdrawal symptoms (response range: 0=not at all, 10=very much).
Intervention acceptability | From baseline to 24-week (i.e., 6-month) follow-up
  Responding to EMA on 25%, 50%, and 75% of days will indicate a low, medium, and high level of acceptability, respectively. An adapted version of a message fatigue measure and a scale of intervention engagement will be used with a response greater than 3 (1 to 5 scales) on each item representing at least some satisfaction with treatment and will serve as the benchmark for acceptability.
Intervention feasibility | From baseline to 24-week (i.e., 6-month) follow-up
  Feasibility benchmarks are assessed continually thoughout the study, beginning with the recruitment rate of eligible participants (≥50% of potential participants) and continuing as quantified by retention at 4 weeks (≥75%), 8 weeks (≥65%), and 24 weeks (≥55%). These data are all proportions and are collected as continuous measures of feasibility as quantified by participant engagement.
Medication adherence | From baseline to 24-week (6-month) follow-up
  Medication for opioid use disorder (MOUD) adherence rate is assessed within individuals. Within-subject adherence will be quantified as ≥80% of days taking MOUD. Six-month between-subject retention rates will be classified using the following ranges based on results from prior studies of buprenorphine and methadone adherence. Buprenorphine: 25% or less = low, 25 to 40% = moderate, and 40% or greater = high. Methadone: 40% of less = low, 40 to 50% = moderate, 50% or greater = high.

SECONDARY OUTCOMES:
Mindfulness text intervention engagement | Measured daily for four weeks
  Participants indicate how much they believe the texting helped them engage in valued activities, engage in everyday activities, be mindful, and accept thoughts and situations without judgement (response range: 0=not at all, 10=very much).
Mindfulness | Measured twice daily for four weeks
  Mindfulness will be assessed through a 6-item EMA scale that measures state mindfulness in the past 15 minutes. Responses are made on a 5-point response scale ranging from 1 (not at all) to 5 (very much).
Pain | Measured twice daily for four weeks
  Pain is assessed using a single-item asking participants to rate their current pain compared to their typical pain level. Responses are made on a 10-point response scale ranging from 0 (a lot less than usual) to 10 (a lot more than usual). A response of 5 represents "about the same as usual.
Pain interference | Measured twice daily for four weeks
  Pain interference is assessed using two items assessing interference with what participants are doing and their enjoyment of life. Responses are made on an 11-point response scale ranging from 0 (not at all) to 10 (very much).
Craving | Measured twice daily for four weeks
  Craving is assessed using 3-items asking participants to rate the: strength of their desire, craving, and urge to use opioids on an 11-point response scale ranging from 0 (not at all) to 10 (very much).
Self-efficacy | Measured twice daily for four weeks
  Self-efficacy is assessed using a single item asking participants to rate their confidence in their ability to not use opioids on an 11-point response scale ranging from 0 (not at all) to 10 (very much).
Values | Measured daily for four weeks
  Values are assessed using two-items adapted from the Values Tracker for EMA measuring engaged with actions that contibute to their quality of living and making progress in life areas that matter to participants. Participants respond on an 11-point response scale ranging from 0 (not at all) to 10 (extremely).
Sleep | Measured daily for four weeks
  Sleep is assessed using three-items. Two are adapted from the Pittsburgh Sleep Quality Index (items 4 and 9) and measure hours of actual sleep (from less than 4 hours to 9 or more hours) and sleep quality rating (from very good [1] to very bad [4]). Participants are also asked to rate how rested they feel ranging from very good (1) to very bad (4).

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States